CLINICAL TRIAL: NCT01796613
Title: Safety and Acceptability of Vaginal Rings That Protect Women From Unintended Pregnancy
Acronym: Ring-Plus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Rinda Ubuzima (Unknown); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ITMC0313
Record Dates: First submitted 2013-02-14; First posted 2013-02-22 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal Ring - intermittent regimen (Active Comparator): 3 weeks ring use followed by one week of no ring use to allow menstruation
  Interventions: Device: Vaginal Ring - intermittent regimen
- Vaginal Ring - continuous regimen (Active Comparator): 3 weeks of ring use with no off period. The next ring is immediately inserted after the previous one
  Interventions: Device: Vaginal Ring - continuous regimen

INTERVENTIONS:
Device: Vaginal Ring - intermittent regimen — NuvaRing® used intermittently. Nuvaring is a contraceptive vaginal ring, manufactured by N.V. Organon (a subsidiary of Merck & Co., Inc.,), Oss, the Netherlands. It contains 11.7 mg etonogestrel and 2.7 mg ethinylestradiol. It releases etonogestrel and ethinylestradiol at an average amount of 0.120 mg and 0.015 mg, respectively per 24 hours, over a period of 3 weeks. It is approved since 2001 by most countries within the European Union, and in the United Stated by the FDA.
  Other Names: NuvaRing®: etonogestrel/ethinylestradiol
  Arms: Vaginal Ring - intermittent regimen
Device: Vaginal Ring - continuous regimen — NuvaRing® used continuously. Nuvaring is a contraceptive vaginal ring, manufactured by N.V. Organon (a subsidiary of Merck & Co., Inc.,), Oss, the Netherlands. It contains 11.7 mg etonogestrel and 2.7 mg ethinylestradiol. It releases etonogestrel and ethinylestradiol at an average amount of 0.120 mg and 0.015 mg, respectively per 24 hours, over a period of 3 weeks. It is approved since 2001 by most countries within the European Union, and in the United Stated by the FDA.
  Other Names: NuvaRing®: etonogestrel/ethinylestradiol
  Arms: Vaginal Ring - continuous regimen

SUMMARY:
The study is a multidisciplinary research project and has two main aims:

1. To determine the safety of a contraceptive vaginal ring (CVR) in women, with an emphasis on its effect on the vaginal microenvironment after different durations of use: the vaginal microbiome, biofilm formation on epithelial cells and rings, inflammation and immune activation in the vagina
2. To investigate the feasibility, acceptability and adherence to vaginal ring use in Rwandan women, including attitudes towards a future multi-purpose vaginal ring for prevention of both pregnancy and sexually transmitted infections (STI).

DETAILED DESCRIPTION:
1. An integrated study design

   This clinical study combines a clinical safety evaluation of the contraceptive vaginal ring (CVR) with social science research on acceptability and adherence of ring use in Rwandan women.

   The clinical part of the study assesses the general safety of the contraceptive ring including the effect on the vaginal microbiome, genitourinary symptoms and signs and clinical adverse events. In addition the clinical part of the study aims to understand better the possible biofilm formation and to explore the impact of the ring on the microbiome and inflammation in the vagina.

   The social science component consists of a combination of a mixed-methods research including In-depth Interviews (IDIs), Focus Group Discussions (FGDs), questionnaires, and (if funding permits) audio computer-assisted self-interviewing (ACASI).
2. Clinical study design

This is an open label single-centre cohort study with the NuvaRing®. A total of 120 Human Immunodeficiency Virus(HIV)-negative women will be randomized to an intermittent regimen or a continuous regimen of ring use and will be followed for maximum 14 weeks, to determine general safety of the ring in the African context, and to determine differences in the vaginal microbiome and vaginal inflammation before and after use of a contraceptive vaginal ring (CVR). Qualitative research for the social science component will be performed to address the acceptability and adherence of intermittent or continuous CVR use in more depth.

Women will be randomized into two study groups: 60 intermittent users in group A and 60 continuous users in group B. Both groups will use the NuvaRing®. Women in group A (the intermittent users) will use each CVR for 3 weeks followed by one week of no ring use to allow menstruation. Women in group B (the continuous users) will use each ring for 3 weeks, with the next ring being inserted immediately after the previous one and no off period in between [4]. The total duration from enrolment to the last study visit is maximum 14 weeks. The screening process will be a maximum of 6 weeks.

As noticed above, the study will include also a social sciences component, aimed at assessing the level of acceptability and reported adherence to intermittent and continuous Contraceptive Vaginal Rings (CVRs) use in women in Rwanda; at identifying and describe the context specific attitudes and beliefs regarding family, family planning, and gendered norms; at exploring the women's beliefs and expectations regarding future potential use of a multi-purpose ring (contraception and Human Immunodeficiency Virus (HIV) prevention); and at exploring how women and men in Rwanda perceive and experience risk related to unwanted pregnancy and Human Immunodeficiency Virus (HIV). This part of the study will result in qualitative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent/assent, according to national guidelines
* Female who self-reports to be sexually active (meaning at least one penetrative vaginal coital act per month for the last 3 months prior to screening)
* Between 18 to 35 years old, inclusive
* Currently in good physical and mental health
* Interested in initiating hormonal contraception
* Able and willing to participate in the study as required by the protocol, this includes willing to undergo HIV testing and use a NuvaRing®
* HIV negative at screening as confirmed by rapid HIV testing

Exclusion Criteria:

* Currently using a modern contraceptive method other than barrier methods
* Use of a hormonal contraceptive method in the three months prior to the screening visit
* Currently using antimicrobial medication
* Pregnant on urine pregnancy test
* History of cardiovascular disease
* History of hysterectomy or genital tract surgery (including cervical polypectomy, dilatation and curettage, hysteroscopy, or laparoscopy) in the three months prior to the screening visit
* History of complications with hormonal contraception or with contra indications for the use of hormonal contraceptives such as:

  * History or known predisposition for venous thrombosis
  * History of migraine with focal neurological symptoms
  * Diabetes mellitus with vascular involvement
  * History of pancreatitis or severe hepatic disease
  * Known or suspected hypersensitivity to any of the excipients of NuvaRing®
* History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding, incontinence or urge incontinence, diagnosed chronic and/or recurrent vulvovaginal candidiasis, urethral obstruction
* Participating in other clinical studies involving investigational products
* Currently breastfeeding
* Currently a smoker

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
vaginal bacterial counts | 5 months
  Changes from baseline (pre-ring use) in vaginal bacterial counts and in the absence/presence of bacterial vaginosis-related bacteria as measured with quantitative real time polymerase chain reaction (PCR).

SECONDARY OUTCOMES:
Incidence of adverse and serious adverse experiences | 5 months
  Incidence of self-reported vaginal symptoms and clinician-observed signs Incidence of bacterial vaginosis. The numbers of women prematurely withdrawing from the study or discontinuing ring use.
  Incidence of adverse and serious adverse experiences . The numbers of incident sexually transmitted infections (STIs) and candidiasis. Nugent scores and Ison & Hay grading of the vaginal flora.
Changes in phenotype of bacterial vaginosis-related bacteria | 5 months
  Changes in phenotype of bacterial vaginosis-related bacteria, specifically:
  * Presence of dispersed forms of bacteria;
  * Presence of adhesive forms of bacteria on epithelial cells.
Presence or absence of a biofilm on the contraceptive vaginal rings (CVRs) | 5 months
  Presence or absence of a biofilm on the Contraceptive Vaginal Rings (CVRs) after intermittent or continuous use:
  * Presence of biofilm visualized by crystal violet; Visualization of adherent bacteria using Fluorescence In Situ Microscopy (FISH);
  * Identification of adherent bacteria (including but not limited to Lactobacilli sp., G. vaginalis, A. vaginae).
Changes in inflammatory cytokines concentrations in Cervicovaginal lavage (CVLs) | 5 months
  Changes in inflammatory cytokines concentrations in Cervicovaginal lavage (CVLs) as measured by Luminex technology. The cytokines analyzed include, but are not limited to Interleukine-1, Interleukine-6, Interleukine-8, Interleukine-10. All samples that are showing elevated cytokine levels, as well as an equal number of controls not showing elevated cytokine levels, will be tested further for the presence of proteins involved in inflammatory pathways.

CONTACTS AND LOCATIONS:
Overall Officials: Tania Crucitti, PhD, Principal Investigator — Institute of Tropical Medicine, Belgium
Locations (1):
- Rinda Ubuzima, Kigali, Rwanda

REFERENCES:
- [Derived] Hardy L, Jespers V, Abdellati S, De Baetselier I, Mwambarangwe L, Musengamana V, van de Wijgert J, Vaneechoutte M, Crucitti T. A fruitful alliance: the synergy between Atopobium vaginae and Gardnerella vaginalis in bacterial vaginosis-associated biofilm. Sex Transm Infect. 2016 Nov;92(7):487-491. doi: 10.1136/sextrans-2015-052475. Epub 2016 Mar 10. PMID 26965870
- [Derived] Schurmans C, De Baetselier I, Kestelyn E, Jespers V, Delvaux T, Agaba SK, van Loen H, Menten J, van de Wijgert J, Crucitti T; RING PLUS study group. The ring plus project: safety and acceptability of vaginal rings that protect women from unintended pregnancy. BMC Public Health. 2015 Apr 10;15:348. doi: 10.1186/s12889-015-1680-y. PMID 25880636